CLINICAL TRIAL: NCT03784989
Title: A Multi-Centre Post Market Clinical Follow-up Study Evaluating Performance and Safety of the SenSura® Mio Kids Device in Subjects With a Stoma
Brief Title: Post Market Clinical Follow-up Study Evaluating Performance and Safety of the SenSura® Mio Kids Device
Status: Withdrawn | Type: Observational
Why Stopped: Lack of recruitment
Sponsor: Coloplast A/S (Industry)
Collaborators: Children's National Research Institute (Other); Driscoll Children's Hospital (Other); IWK Health Centre (Other)
Responsible Party: Sponsor
Other Study IDs: CP281
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Stoma Ileostomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a post market clinical follow-up study and devices will carry the CE mark once the study is initiated.

The investigational device is SenSura® Mio Kids, which is a flat ostomy device. The device is comprised by a baseplate connected to a bag. The coupling between baseplate and bag can be either welded together, referred to as a 1-piece (1P) system, or assembled as separate parts, referred to as a 2-piece (2P) system.

DETAILED DESCRIPTION:
The purpose of this research is to gather more information about how well the SenSura® Mio Kids ostomy device works, and how safe it is. This device has already been studied and approved to be used in the United States. It has a European CE-mark, which means it has met European health and safety requirements. SenSura® Mio Kids is a flat ostomy device that is made to be used for kids from 6 months up to 4 years of age.

The reason for this study is to find out how well the new SenSura® Mio Kids device works compared to the standard of care device. We can learn about this by asking people who have used it about how well it worked and how comfortable it was.

The Investigator/study nurse will decide whether the subject would benefit from switching to SenSura® Mio Kids and if so, the subject will be invited to take part in the study. The study design is observational. That means that the ostomy device, and the skin around the stoma, will be observed while receiving the stoma care they normally would. This study design will help the researchers see how well the device works when it is used in the usual way, and makes it easier for the people who are participating in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Have a colostomy, ileostomy, urostomy, loop stoma, or two stomas placed closely together
2. Have given written informed consent (the legal authorized representative of the subject)
3. Group 1 subjects should use a competitor device

Exclusion Criteria:

1) Are currently suffering from peristomal skin problems i.e. bleeding and/or broken skin (as-sessed by the investigator)

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The population in this study are subjects from the age of 6 months (calculated from term age meaning 40 gestational weeks) to 4 years either with a colo-, ileo- or urostomy or a loop stoma, or two stomas placed closely together. Subjects can participate in the PMCF study if they fulfill the in-/exclusion criteria as listed in the tables below. However, the per protocol population only include 30 subjects as needed for the compara-tive performance evaluation (Group 1), and these subjects must fulfill inclusion criteria no. 3 (subjects should use a competitor device).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Median wear time | 2-3 weeks
  of 8 baseplate changes

CONTACTS AND LOCATIONS:
Locations (1):
- Driscoll Childrens Hospital, Corpus Christi, Texas, United States